CLINICAL TRIAL: NCT01626404
Title: Screening for Advanced Heart Failure Treatment (SEE-HF)
Acronym: SEE-HF
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Thoratec Europe Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: TC-060112
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Advanced Heart Failure; CRT and/or ICD
Keywords: Thoratec Corporation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients enrolled: All patients enrolled in the study

SUMMARY:
Advanced heart failure therapy (heart transplantation or LVAD) is underutilized and patients are underserved. The purpose of this prospective, observational study is to obtain multi-center data on the proportion of patients with CRT and/or ICD who are candidates for advanced heart failure treatment and obtain insights into patient and physician decisions regarding referral for advanced heart failure therapy.

ELIGIBILITY:
Inclusion Criteria:

* CRT and or ICD device in place.
* NYHA class III - IV heart failure
* EF </= 40%
* Patient is an out-patient
* Patient is on optimal medical management as tolerated and as defined by primary care physician.
* Patient has signed an informed consent for data collection.

Exclusion Criteria:

* Age <18 years or >80 years
* CRT device that has been implanted < 3 months prior to enrollment
* Coronary revascularization within 3 months prior to enrollment
* Patient only has ICD but has CRT planned
* Non-cardiac disease resulting in life expectancy < 2 yrs
* Patient is hospitalized or will be hospitalized at this time
* Known diagnosis of dementia
* Patient is currently on dialysis
* Oxygen dependent lung disease
* Previously or currently treated with LVAD or heart transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with CRT and/or ICD, EF </= 40% and in NYHA III-IV
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2012-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients | 12 months
  Proportion of heart failure patients followed in outpatient clinic that are NYHA III-IV with LVEF </= 40% and a CRT and/or ICD who have an indication without contraindication for heart transplantationi and/or DT LVAD.

SECONDARY OUTCOMES:
Reasons for non-referral | 12 months
  Assess physician's reasons for non-referral of patients for LVAD/transplant evaluation.
Patient's reasons | 12 months
  Assess patients reasons for declining LVAD/transplant as a treatment option.
Actual and predicted 12 month survival | 12 months
  Assess the actual and predicted 12 month survival (predicted by VO2, the Heart Failure Survival Score (HFSS) and the Seattle Heart Failure Model (SHFM)).
Simple clinical parameters for referral | 12 months
  Identify simple clinical parameters that can be used by physicians to refer patients for LVAD/transplant evaluation at an optimal time.

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Chatterjee, Study Director — Thoratec Europe Limited
Locations (7):
- Rigshospitalet, Copenhagen, Denmark
- CHU of Nantes, Nantes, France
- Germany (2):
  - Hannover Medical Center, Hanover
  - University Clinical Center Tuebingen, Tübingen
- Erasmus Medical Center, Rotterdam, Netherlands
- Karolinska University Hospital, Stockholm, Sweden
- University Hospital of South Manchester NHS Trust, Manchester, United Kingdom